CLINICAL TRIAL: NCT00994123
Title: A Phase 1-2 Trial of MM-121 in Combination With Erlotinib in Three Groups of Patients With Non-Small Cell Lung Cancer
Brief Title: A Study of MM-121 Combination Therapy in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-01-101
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer; NSCLC; Advanced Non-Small Cell Lung Cancer; Metastatic Non-Small Cell Lung Cancer; Lung Cancer; Erlotinib; Tarceva; MM-121; ErbB3; Her3; Epidermal Growth Factor Receptor; anti-ErbB3 human monoclonal antibody; ErbB3 antagonist
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Lethal Congenital Contracture Syndrome 2 | interventions — seribantumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1: Dose-Escalation (Experimental): Escalating doses of MM-121 (QOW IV) and erlotinib (daily PO)
  Interventions: Drug: MM-121; Drug: Erlotinib
- Phase 2: Control (Active Comparator): Erlotinib (daily)
  Interventions: Drug: Erlotinib
- Phase 2: Treatment (Experimental): MM-121 (QOW IV) and erlotinib (daily PO)
  Interventions: Drug: MM-121; Drug: Erlotinib

INTERVENTIONS:
Drug: MM-121 — MM-121 (SAR256212) = intravenous solution
  Other Names: SAR256212
  Arms: Phase 1: Dose-Escalation; Phase 2: Treatment
Drug: Erlotinib — erlotinib = daily oral tablet
  Other Names: Tarceva

SUMMARY:
A Phase 1-2 study of MM-121 in combination with standard therapy for non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Phase 1: Patients with Non-Small Cell Lung Cancer (NSCLC) may be enrolled to evaluate the safety, tolerability and recommended Phase 2 dose of MM-121 in combination with standard therapy.

Phase 2: Patients with Non-Small Cell Lung Cancer (NSCLC) may be enrolled to estimate the progression-free survival of the MM-121 + standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic non-small cell lung cancer.
* Patients must be >/= 18 years of age.
* Patients must have adequate Performance Status (PS) as measured by ECOG and adequate end organ function.

Exclusion Criteria:

* Patients with a recent history (within 5 years) of another malignancy.
* Patients who are pregnant or nursing.
* Patients with clinically significant heart failure.
* Patients with clinically significant eye or gastrointestinal abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Moyo, MD, Study Director — Merrimack Pharmaceuticals
Locations (37):
- United States (19):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Loma Linda, California
  - Sacramento, California
  - San Francisco, California
  - Aurora, Colorado
  - Tampa, Florida
  - Atlanta, Georgia
  - Lafayette, Indiana
  - Boston, Massachusetts
  - St Louis, Missouri
  - Buffalo, New York
  - New York, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
- Canada (3):
  - Edmonton, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (6):
  - Heidelberg, Mannheim
  - Bad Berka
  - Frankfurt
  - Heidelberg
  - Lungenklinik
  - Ulm
- South Korea (2):
  - Seoul, Gangnam-gu
  - Seoul, Seodaemun-gu
- Spain (3):
  - Barcelona
  - Madrid
  - Málaga
- Taiwan (4):
  - Guishan, Taoyuan County
  - Taichung
  - Tainan
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: MM-121 + Erlotinib: Escalating doses of MM-121 and erlotinib
- Phase 2: MM-121 + Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  MM-121 every other week at a dose of 20 mg/kg IV in combination with daily 100 mg erlotinib p.o.
- Phase 2: Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  daily 150 mg erlotinib p.o. alone
Period: Overall Study
Arm/Group | Phase 1: MM-121 + Erlotinib | Phase 2: MM-121 + Erlotinib | Phase 2: Erlotinib
Started | 33 | 85 | 44
Completed | 33 | 85 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ph 1: Patients with NSCLC Ph 2:Patients whose tumors are wild-type for EGFR and who have not received prior EGFR TKI targeted therapy.
Groups:
- Phase 1: MM-121 + Erlotinib: Escalating doses of MM-121 + Erlotinib in patients with NSCLC
- Total: Total of all reporting groups
Arm/Group | Phase 1: MM-121 + Erlotinib | Phase 2: MM-121 + Erlotinib | Phase 2: Erlotinib | Total
Number analyzed (Participants) | 33 | 85 | 44 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.12) | 62.9 (10.74) | 63.9 (10.16) | 63.2 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 35 | 17 | 69
  Male | 16 | 50 | 27 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 31 | 82 | 43 | 156
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 7
  White | 31 | 74 | 36 | 141
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: To Determine the Recommended Phase 2 Dose of the MM-121 + Erlotinib Combination Based Upon Either the Maximum Tolerated Dose (MTD) or the Maximum Feasible Dose of the Combination in Patients With NSCLC.
Description: To establish the safety of escalating doses of MM-121 in combination with erlotinib in order to determine the recommended phase 2 dose of the combination for the second part of the study. Dose-escalation conducted using standard 3+3 model to determine maximum tolerated dose. Reports of Dose-Limiting Toxicities (DLTs) were assessed to determine the MTD.
Time Frame: From date of first dose to 30 days after termination, the longest 175 weeks
Measure: Number; unit: participants reporting DLTs
Groups:
- Cohort 1: MM-121 6 mk/kg (Q2W IV) and 100 mg erlotinib (daily PO)
- Cohort 2: 6 mg/kg MM-121 Q2W + 150 mg erlotinib (daily PO)
- Cohort 3: MM-121 12 mg/kg (Q2W IV) + 100 mg erlotinib (daily PO)
- Cohort 4: MM-121 12 mg/kg (Q2W IV) + 150 mg erlotinib (PO daily)
- Cohort 5: MM-121 20 mg/kg (weekly IV) + erlotinib 100 mg (PO daily)
- Cohort 6: MM-121 20 mg/kg (Q2W IV) + erlotinib 100 mg (PO daily)
- Cohort 7: MM-121 20 mg/kg (Q3W IV) + erlotinib 100 mg (PO daily)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 1 | 3 | 6 | 3 | 6 | 8 | 6
participants reporting DLTs | 0 | 0 | 1 | 1 | 1 | 0 | 0

2. Primary Outcome: Phase 1: Determine the Maximum Tolerated Dose Dependent on Reports of Dose-limiting Toxicities
Description: Using a 3+3 dose escalation model, the maximum tolerated dose was determined by assessing dose-limiting toxicities in each cohort. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in the expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs.
  The determined MTD was used as the recommended Phase 2 dose.
Time Frame: From date of first dose to 30 days after termination, the longest 175 weeks
Population: All participants treated in the Phase 1 dose-escalation portion of the study
Measure: Number; unit: dose level of MTD
Groups:
- Phase 1: All Participants: All participants in the dose escalation portion of the Phase 1
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 33
dose level of MTD | NA — Maximum tolerated dose was not reached. Recommended Phase 2 Dose (MM-121 mg/kg IV Q2W + erlotinib 100 mg PO daily) was selected based on Investigator agreement on safety profile and PK parameters.

3. Primary Outcome: Phase 2: Progression-free Survival of the MM-121 + Erlotinib Combination
Description: This was a time-to-event measure using Progression-Free Survival (PFS) comparing MM-121 + erlotinib vs.erlotinib alone. Progression of disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions". Progression free survival was defined as the number of weeks from the date of randomization to the date of death or progression. If neither death nor progression was observed during the study, PFS data was censored at the last non-progressive disease valid tumor assessment unless the patient was discontinued due to symptomatic deterioration. If this occurred, the patient was counted as having progressive disease (PD).
Time Frame: Time from first dose to date of progression, with a median of 8.1 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- MM-121 + Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  MM-121 every other week at a dose of 20 mg/kg IV in combination with daily 100 mg erlotinib p.o.
- Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  daily 150 mg erlotinib p.o. alone
Arm/Group | MM-121 + Erlotinib | Erlotinib
Number analyzed (Participants) | 85 | 44
weeks | 8.1 [7.7 to 8.9] | 7.7 [7.1 to 8.1]

4. Post Hoc Outcome: To Explore the Utility of an EGFR Family Receptor-ligand (Heregulin, HRG) as a Predictor of Response to MM-121 and /or Erlotinib in Formalin Fixed (FFPE) Tumor Samples
Description: Tumor tissue samples were obtained from patients prior to enrollment. Samples were analyzed using RNA-ISH for the expression of the biomarker, heregulin. Progression-free survival was assessed using RECIST v 1.1 to determine whether patients whose tumors express HRG have a lower PFS than those whose tumors do not express HRG, and to assess whether the addition of MM-121 to erlotinib can increase PFS in HRG-high patients.
Time Frame: Time from first dose to date of progression, with a median of 8.1 weeks
Population: Patients with available tissue for heregulin testing
Measure: Median (95% Confidence Interval); unit: months PFS
Groups:
- HRG High: MM-121 + Erlotinib; HRG Low: MM-121 + Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  MM-121 every other week at a dose of 20 mg/kg IV in combination with daily 100 mg erlotinib p.o.
- HRG High: Erlotinib; HRG Low: Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  daily 150 mg erlotinib p.o. alone
Arm/Group | HRG High: MM-121 + Erlotinib | HRG High: Erlotinib | HRG Low: Erlotinib | HRG Low: MM-121 + Erlotinib
Number analyzed (Participants) | 23 | 13 | 12 | 20
months PFS | 1.9 [1.7 to 4] | 1.7 [1 to NA] — Upper bound was not evaluable due to too few events | 2.3 [1.7 to NA] — Upper bound was not evaluable due to too few events | 1.6 [1.4 to 1.9]
Statistical Analysis 1: Comparison: HRG High: MM-121 + Erlotinib vs HRG High: Erlotinib; Test type: Superiority or Other; p = 0.008, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.16 to 0.76]
Statistical Analysis 2: Comparison: HRG Low: Erlotinib vs HRG Low: MM-121 + Erlotinib; Test type: Superiority or Other; p = 0.059, Log Rank; Hazard Ratio (HR) = 2.15, 95% CI 2-sided [0.97 to 4.76]

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination.
Groups:
- Ph 2: MM-121 + Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  MM-121 every other week at a dose of 20 mg/kg IV in combination with daily 100 mg erlotinib p.o.
- Ph 2: Erlotinib: EGFR wild-type, EGFR-TKI naive patients randomized to receive:
  daily 150 mg erlotinib p.o. alone
- Ph 1: MM-121 + Erlotinib: Escalating Doses of MM-121 + erlotinib
Arm/Group | Ph 2: MM-121 + Erlotinib | Ph 2: Erlotinib | Ph 1: MM-121 + Erlotinib
Serious Adverse Events (participants affected / at risk) | 40/85 | 18/44 | 16/33
Other Adverse Events (participants affected / at risk) | 85/85 | 44/44 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ph 2: MM-121 + Erlotinib (N=85) | Ph 2: Erlotinib (N=44) | Ph 1: MM-121 + Erlotinib (N=33)
Disease Progression (General disorders) | 14 | 3 | 1
Chest Pain (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Gait Disturbance (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Klebsiella Infection (Infections and infestations) | 0 | 1 | 0
Localized Infection (Infections and infestations) | 1 | 0 | 0
Scrotal Infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary Tumor Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pericardial effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1 | 0
Intracardiac Thrombus (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 2
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Complex Partial Seizures (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
General Physical Condition Abnormal (Investigations) | 1 | 0 | 0
International Normalized Ratio Increased (Investigations) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Dermatitis Acneform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hemorrhage (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Venous Occlusion (Vascular disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ph 2: MM-121 + Erlotinib (N=85) | Ph 2: Erlotinib (N=44) | Ph 1: MM-121 + Erlotinib (N=33)
Rash (Skin and subcutaneous tissue disorders) | 46 | 21 | 15
Dry Skin (Skin and subcutaneous tissue disorders) | 28 | 11 | 11
Dermatitis Acneform (Skin and subcutaneous tissue disorders) | 14 | 12 | 12
Pruritis (Skin and subcutaneous tissue disorders) | 10 | 10 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 4 | 3
Palmar-Plantar Erythrodysasthesia Syndrome (Skin and subcutaneous tissue disorders) | 4 | 3 | 3
Skin Disorder (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 0 | 3
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 3 | 0 | 4
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 59 | 27 | 27
Nausea (Gastrointestinal disorders) | 29 | 14 | 9
Vomiting (Gastrointestinal disorders) | 19 | 11 | 8
Stomatitis (Gastrointestinal disorders) | 20 | 5 | 7
Constipation (Gastrointestinal disorders) | 10 | 7 | 6
Abdominal Pain (Gastrointestinal disorders) | 5 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 4
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 2 | 2
CHEILITIS (Gastrointestinal disorders) | 0 | 0 | 2
DRY MOUTH (Gastrointestinal disorders) | 3 | 0 | 2
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 31 | 13 | 21
Disease Progression (General disorders) | 14 | 3 | 1
Asthenia (General disorders) | 7 | 6 | 3
Pyrexia (General disorders) | 6 | 7 | 1
Mucosal Inflammation (General disorders) | 9 | 3 | 7
Peripheral Edema (General disorders) | 4 | 3 | 6
Early Satiety (General disorders) | 1 | 0 | 7
Pain (General disorders) | 0 | 0 | 4
Chills (General disorders) | 4 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 9 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 6 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 6
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 37 | 16 | 11
Hypokalemia (Metabolism and nutrition disorders) | 14 | 3 | 8
Dehydration (Metabolism and nutrition disorders) | 7 | 5 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 3 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 3
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 3
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 2
Weight Decreased (Investigations) | 27 | 11 | 9
Blood Creatinine Increased (Investigations) | 7 | 3 | 2
Aspartate Aminotransferase Increased (Investigations) | 6 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 6 | 1 | 1
Blood Magnesium Decreased (Investigations) | 6 | 0 | 0
Blook Alkaline Phosphatase Increased (Investigations) | 5 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 3
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 | 0 | 2
Breath Sounds Abnormal (Investigations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 6 | 6 | 2
Paronychia (Infections and infestations) | 9 | 2 | 7
Urinary Tract Infection (Infections and infestations) | 4 | 4 | 9
Nasopharyngitis (Infections and infestations) | 3 | 3 | 0
CANDIDIASIS (Infections and infestations) | 0 | 0 | 3
FUNGAL SKIN INFECTION (Infections and infestations) | 2 | 1 | 3
UPPER RESPIRATORY TRACT (Infections and infestations) | 4 | 1 | 3
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 3
NAIL INFECTION (Infections and infestations) | 1 | 0 | 2
Oral Herpes (Infections and infestations) | 3 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 4 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 11 | 8 | 4
Dysgeusia (Nervous system disorders) | 14 | 1 | 6
Headache (Nervous system disorders) | 7 | 3 | 3
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 1 | 3
AMNESIA (Nervous system disorders) | 0 | 0 | 2
PARAESTHESIA (Nervous system disorders) | 3 | 2 | 2
SYNCOPE (Nervous system disorders) | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 8 | 2 | 4
Depression (Psychiatric disorders) | 5 | 3 | 2
Insomnia (Psychiatric disorders) | 5 | 1 | 12
Confusional State (Psychiatric disorders) | 1 | 3 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 9 | 4 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 0 | 5
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 2
NOCTURIA (Renal and urinary disorders) | 1 | 0 | 2
PROTEINURIA (Renal and urinary disorders) | 1 | 0 | 2
CONJUNCTIVITIS (Eye disorders) | 3 | 0 | 4
EYE PAIN (Eye disorders) | 1 | 0 | 2
EYE PRURITUS (Eye disorders) | 0 | 0 | 2
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 2
TACHYCARDIA (Cardiac disorders) | 1 | 1 | 3
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 0 | 2
HYPERTENSION (Vascular disorders) | 1 | 1 | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 2
hyperbilirubinemia (Hepatobiliary disorders) | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less